CLINICAL TRIAL: NCT00598208
Title: A Phase 2, Open Label, Randomized Trial to Investigate the Dose-Response Relationship of a Single Injection of Org 36286 (Corifollitropin Alfa) to Initiate Multiple Follicular Growth in a Controlled Ovarian Hyperstimulation Protocol for IVF or ICSI.
Brief Title: A Phase 2, Trial to Investigate the Dose-Response Relationship of a Single Injection of Org 36286 (Corifollitropin Alfa) to Initiate Multiple Follicular Growth in a Controlled Ovarian (Study 38826)(P06055)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06055; 38826
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Fertilization
Keywords: In-vitro fertilization
MeSH Terms: interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 60 µg Org 36286 (corifollitropin alfa)
  Interventions: Drug: corifollitropin alfa
- 2 (Experimental): 120 µg Org 36286 (corifollitropin alfa)
  Interventions: Drug: corifollitropin alfa
- 3 (Experimental): 180 µg Org 36286 (corifollitropin alfa)
  Interventions: Drug: corifollitropin alfa
- 4 (Active Comparator): Follitropin beta injection
  Interventions: Drug: Follitropin beta injection

INTERVENTIONS:
Drug: corifollitropin alfa — On Cycle Day 2, a single injection of 60 μg, 120 μg, or 180 μg Org 36286 was administered. One week later (Treatment Day 8), treatment was continued with a fixed daily subcutaneous (SC) dose of 150 IU Puregon® up to and including the Day of hCG. Orgalutran® (0.25 mg) was administered once daily SC starting on Treatment Day 5 and up to and including the Day of hCG. The maximum total treatment duration was 19 days.
  Other Names: Org 36286
  Arms: 1; 2; 3
Drug: Follitropin beta injection — Starting on Cycle Day 2, a fixed daily dose of 150 IU Puregon® SC was administered for the entire stimulation period up to and including the Day of hCG. Orgalutran® (0.25 mg) was administered once daily SC starting on Treatment Day 5 and given up to and including the day of hCG. The maximum total treatment duration was 19 days.
  Other Names: Follistim®; Puregon®
  Arms: 4

SUMMARY:
The primary objective of this trial is to investigate the dose -response relationship of a single injection of Org 38286 to initiate multifollicular growth for the first seven days in a controlled ovarian hyperstimulation (COH) protocol for IVF or ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Females of couples with an indication for COH and IVF or ICSI;
* >=18 and <=39 years of age at the time of signing informed consent;
* BMI >=18 and <=29 kg/m^2;
* Normal menstrual cycle length: 24-35 days;
* Ejaculatory sperm (use of donated and/or frozen sperm is allowed);
* Willing and able to sign informed consent.

Exclusion Criteria:

* History of/or any current (treated) endocrine abnormality;
* History of ovarian hyperstimulation syndrome (OHSS);
* History of/or current polycystic ovary syndrome (PCOS) or current polycystic ovaries according to USS (at least 10 follicles of 2-8 mm in each ovary);
* More than three unsuccessful COH cycles since the last established ongoing pregnancy (if applicable);
* History of non- or low ovarian response to FSH/hMG treatment;
* Any clinically relevant hormone value outside the reference range during the early follicular phase (menstrual cycle day 2-7) as measured by the local laboratory (FSH, LH, E2, P, total T, TSH and prolactin):
* Any clinically relevant abnormal laboratory value;
* Less than 2 ovaries;
* Any ovarian and/or abdominal abnormality interfering with ultrasound examination;
* Contraindications for the use of gonadotropins (e.g. tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, ovarian cysts);
* Epilepsy, diabetes, cardiovascular, gastro-intestinal, hepatic, renal, pulmonary, or abdominal disease;
* History of presence of alcohol or drug abuse within 12 months prior to signing informed consent;
* Previous use of Org 36286;
* Use of hormonal preparations within 1 month prior to randomization;
* Hypersensitivity to Org 32489 (Puregon®) and/or Org 37462 (Orgalutran®) and/or Pregnyl® or any of their components;
* Administration of investigational drugs within three months prior to signing informed consent.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 325 (Actual)
Dates: Start 2003-05-19 (Actual); Primary Completion 2004-03-15 (Actual); Study Completion 2004-03-15 (Actual)

PRIMARY OUTCOMES:
Number of cumulus-oocyte-complexes retrieved | 1 cycle

SECONDARY OUTCOMES:
Treatment failure rate | 1 cycle

REFERENCES:
- [Derived] Zandvliet AS, Prohn M, de Greef R, van Aarle F, McCrary Sisk C, Stegmann BJ. Impact of patient characteristics on the pharmacokinetics of corifollitropin alfa during controlled ovarian stimulation. Br J Clin Pharmacol. 2016 Jul;82(1):74-82. doi: 10.1111/bcp.12939. Epub 2016 May 31. PMID 26991902
- [Derived] Corifollitropin Alfa Dose-finding Study Group. A randomized dose-response trial of a single injection of corifollitropin alfa to sustain multifollicular growth during controlled ovarian stimulation. Hum Reprod. 2008 Nov;23(11):2484-92. doi: 10.1093/humrep/den288. Epub 2008 Aug 6. PMID 18684735